CLINICAL TRIAL: NCT01180855
Title: Effects of Ramelteon (8mg) Alone and in Combination With Multi-Component Behavioral Therapy on Sleep and Circadian Phase in Patients With Chronic Insomnia: A Randomized, Double-Blind, Placebo Controlled Study (Investigator Initiated Study)
Brief Title: Effects of Ramelteon (8mg) Alone and in Combination With Multi-Component Behavioral Therapy on Sleep and Circadian Phase in Patients With Chronic Insomnia
Acronym: CBT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arizona (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Richard R. Bootzin, PhD Professor of Psychology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-046R
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Insomnia
Keywords: Melatonin; Cognitive Behavior Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo pills prepared by Takeda Pharmaceutical.
  Interventions: Drug: Placebo
- Rozerem (Active Comparator): Rozerem 8mg
  Interventions: Drug: Rozerem 8mg
- Rozerem + Multi Component Behavior Therapy (Active Comparator): Rozerem 8mg in combination with 4 small group sessions and 2 phone calls of Multi Component Behavior Therapy.
  Interventions: Other: Rozerem 8mg in combination with Multi Component Behavior Therapy

INTERVENTIONS:
Drug: Placebo — Placebo pill nightly for 42 nights.
  Arms: Placebo
Drug: Rozerem 8mg — Rozerem 8mg pill, nightly for 42 nights
  Arms: Rozerem
Other: Rozerem 8mg in combination with Multi Component Behavior Therapy — Rozerem 8mg pill nightly for 42 nights with 4 sessions and 2 telephone calls of Multi Component Behavior Therapy.
  Arms: Rozerem + Multi Component Behavior Therapy

SUMMARY:
The specific aims of the proposed study are to compare the sleep, daytime functioning, and circadian phase effects of ROZEREMTM (ramelteon/TAK-375) a selective MT1/MT2 melatonin receptor agonist in humans alone and in combination with multi-component behavior therapy (MCBT) in patients with chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Medical and sleep/wake history. During the screening process, participants will receive a physical exam, urine and blood labs, and be interviewed about their medical and sleep/wake history and be asked questions about their present and past habitual sleep/wake schedule and nap times.

  (b) Medication/drug/alcohol use. Participants must have no history of drug or alcohol abuse or dependency, consume no more than 2 alcoholic beverages a day or more than 14 per week, Participants must agree not to consume more than 2 beverages containing caffeine (caffeinated coffee, tea, colas) a day before 2 pm and none after 2 pm.

  (c) Evaluation of Psychiatric/Psychological Suitability. Participants must demonstrate a full understanding of the requirements and demands of the study.

For inclusion/exclusion screening, participants will receive a sleep, medical, physical and psychiatric history examination, one-night of dim light melatonin onset evaluation in the sleep laboratory, one-night of polysomnography, and two weeks of baseline sleep assessment. If during the polysomnography assessment the participant had a respiratory disturbance index (RDI) of 15 or more, the participant would be considered to have met the exclusionary criterion for obstructive sleep apnea. A letter providing feedback of the all night polysomnography assessment will be sent to all participants.

Individuals with a history of psychiatric illnesses or psychiatric disorders will be excluded, such as but not limited to, alcoholism, drug dependency, mood disorders; schizophrenic disorders, anxiety disorders; personality disorders. Finally, individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressants, neuroleptic medications or major tranquilizers will be excluded from study. However, a personal history of limited prior counseling or psychotherapy (e.g., for adjustment reactions) will not be exclusionary. Individuals who have been treated for insomnia within the past six months will be excluded.

Exclusion Criteria:

* Exclusion criteria include diagnosis or treatment of other sleep disorders such as obstructive sleep apnea, narcolepsy, sleep walking, and periodic limb movement disorders. Participants with a history of night work in the preceding 6 months or transmeridian travel (across >3 time zones) in the last 1 month prior to the study will be excluded.

Use of psychotropic, hypnotic medications known to affect sleep or contraindicated for use with ramelteon, or over-the-counter analgesics that contain caffeine, or herbal supplements, including products with herbs, melatonin, or St. John's Wort.

Substance use will be determined by self-report and urine toxicology during the screening visit. Women who are pregnant or are planning on becoming pregnant will be excluded from the study. Female participants will be given a pregnancy test during the screening process.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Sleep Onset Latency | Baseline, Post treatment, 3 month follow up
  Daily assessment of sleep and daytime functioning (daily voice mail sleep diary and actigraphy) for 10 weeks: 2 weeks prior to and after treatment and during the 6 week treatment period. The primary sleep outcomes will be improvement in sleep onset latency (SOL) and total sleep time (TST).

SECONDARY OUTCOMES:
Dim Light Melatonin Onset | Baseline, post treatment
  Assessment of circadian melatonin phase 2 weeks prior to and 2 weeks after treatment(dim light melatonin onset-DLMO, 2 weeks prior to treatment and 2 weeks post treatment assessment of quality of life (SF-36) and sleep quality (Pittsburgh Sleep Quality Index-PSQI), 2 weeks prior to treatment and 2 weeks post treatmemnt daily assessment of daytime functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Bootzin, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Sleep Research Laboratory, Tucson, Arizona, United States